CLINICAL TRIAL: NCT01360021
Title: A 12-week, Double-blind, Randomized, Multi-centre, Parallel-group Study Evaluating the Efficacy Safety, and Patient Use (User Study) of Symbicort® (Budesonide/Formoterol) Breath Actuated Metered Dose Inhaler (BA MDI) 2x160/4.5 μg Twice Daily Compared With Symbicort (Budesonide/Formoterol) AC (Actuation Counter) pMDI® 2x160/4.5 μg Twice Daily and Budesonide AC pMDI 2x160 μg Twice Daily in Adult and Adolescent Asthmatics
Brief Title: New Breath Actuated MDI Symbicort Compared to Symbicort pMDI and Budesonide pMDI for 12 Weeks Twice a Day
Acronym: BAI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D589OC00003
Record Dates: First submitted 2011-05-19; First posted 2011-05-25 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 Symbicort/inhaler (Active Comparator): Symbicort BA MDI 2x160/4.5 μg twice daily
  Interventions: Drug: Symbicort
- Symbicort/inhaler (Active Comparator): Symbicort AC pDMI 2x160/4.5 μg twice daily
  Interventions: Drug: Symbicort
- Budesonide/inhaler (Active Comparator): Budesonide AC pMDI 2x160 μg twice daily
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Symbicort — Breath actuated metered dose inhaler
  Arms: 1 Symbicort/inhaler
Drug: Symbicort — Actuation counter pressured metered dose inhaler
  Arms: Symbicort/inhaler
Drug: Budesonide — Actuation counter pressured metered dose inhaler
  Arms: Budesonide/inhaler

SUMMARY:
This is a comparison of the efficacy of the Symbicort breath actuated dose inhaler to the Symbicort pressured meter dose inhaler after 12 weeks of a twice a day dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 12 years and above
* Clinical diagnosis of asthma according to the American Thoracic Society definition at least 6 months
* Pre-bronchodilator FEV1 ≥ 45% and ≤ 85% of predicted normal
* Patients with reversible airway obstruction
* Documented daily use of inhaled corticosteroids for ≥ 3 months

Exclusion Criteria:

* History of life-threatening asthma, defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures during the 2 years prior to Visit 2
* Hospitalized during previous 6 months for asthma
* Required emergency treatment more than once during previous 6 months for an asthma-related condition
* Intake of oral, rectal or parenteral glucocorticosteroid within 30 days of enrolment
* Respiratory infection affecting the asthma within 30 days

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goran Eckerwall, MD, Study Director — AstraZeneca R&D, Mölndal
Locations (41):
- United States (31):
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Rancho Mirage, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Tallahassee, Florida
  - Research Site, Savannah, Georgia
  - Research Site, River Forest, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Wheaton, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Columbia, Missouri
  - Research Site, Rolla, Missouri
  - Research Site, Skillman, New Jersey
  - Research Site, North Syracuse, New York
  - Research Site, Rochester, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Collegeville, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Tacoma, Washington
  - Research Site, Greenfield, Wisconsin
  - Research Site, Madison, Wisconsin
- Bulgaria (4):
  - Research Site, Rousse, Bulgaria
  - Research Site, Sevlievo, Bulgaria
  - Research Site, Sofia, Bulgaria
  - Research Site, Varna, Bulgaria
- Hungary (4):
  - Research Site, Balassagyarmat, Hungary
  - Research Site, Budapest, Hungary
  - Research Site, Salgótarján, Hungary
  - Research Site, Százhalombatta, Hungary
- Russia (2):
  - Research Site, Moscow, Russia
  - Research Site, Yekaterinburg, Russia

REFERENCES:
- [Derived] Murphy KR, Dhand R, Trudo F, Uryniak T, Aggarwal A, Eckerwall G. Therapeutic equivalence of budesonide/formoterol delivered via breath-actuated inhaler vs pMDI. Respir Med. 2015 Feb;109(2):170-9. doi: 10.1016/j.rmed.2014.12.009. Epub 2015 Jan 3. PMID 25596138

RESULTS

PARTICIPANT FLOW:
Groups:
- Symbicort BA MDI: Symbicort BA MDI 2x160/4.5 μg twice daily
- Symbicort pMDI: Symbicort AC pDMI 2x160/4.5 μg twice daily
- Budesonide: Budesonide AC pMDI 2x160 μg twice daily
Period: Overall Study
Arm/Group | Symbicort BA MDI | Symbicort pMDI | Budesonide
Started | 71 (Patients randomized) | 71 (Patients randomized) | 72 (Patients randomized)
Completed | 63 (Patients who completed study) | 67 (Patients who completed study) | 65 (Patients who completed study)
Not Completed | 8 | 4 | 7
Not completed — Eligibility criteria + other | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 2
Not completed — Adverse Event | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All Randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort BA MDI | Symbicort pMDI | Budesonide | Total
Number analyzed (Participants) | 71 | 71 | 72 | 214
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.83 (16.156) | 42.62 (16.873) | 42.72 (14.424) | 42.72 (15.770)
Age, Customized [Number; unit: Participants]
  12 - <18 years | 6 | 8 | 7 | 21
  18 - <65 years | 60 | 56 | 62 | 178
  65 - <75 years | 4 | 4 | 2 | 10
  >= 75 years | 1 | 3 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 47 | 35 | 119
  Male | 34 | 24 | 37 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 9 | 7 | 11 | 27
  White | 57 | 63 | 57 | 177
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Years since asthma diagnosis [Mean (Standard Deviation); unit: Years] | 24.26 (14.891) | 24.12 (15.128) | 24.38 (15.183) | 24.25 (14.998)
% Predicted FEV1 (Visit 2) [Mean (Standard Deviation); unit: %] | 67.27 (10.048) | 65.02 (11.135) | 68.49 (9.924) | 66.93 (10.434)
% Reversibility in FEV1 (Visit 2) [Mean (Standard Deviation); unit: %] — Reversibility is defined as a change of ≥12% in FEV1 from pre-bronchodilator values (for patients ≥12 and <18 years of age), and for patients ≥18 years of age, a change of ≥12% and 200 mL in FEV1 from pre-bronchodilator values. Percent reversibility of FEV1 was calculated as follows: (Post-bronchodilator FEV1 - pre-bronchodilator FEV1)/pre-bronchodilator FEV1 x 100.
  % | 23.93 (15.728) | 28.04 (14.712) | 23.64 (12.692) | 25.20 (14.491)
% Reversibility in FEV1 (Visit 3) [Mean (Standard Deviation); unit: %] | 26.43 (16.662) | 28.22 (16.118) | 24.88 (14.235) | 26.51 (15.692)
Baseline % Predicted FEV1 (Visit 4) [Mean (Standard Deviation); unit: %] | 67.78 (11.059) | 67.31 (10.683) | 68.27 (11.078) | 67.79 (10.898)

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) - Post Dose
Description: Descriptive statistics for post-dose FEV1 (L) by visit; Baseline defined as the last pre-dose value prior to 1st dose of randomized therapy. Trt Avg = Mean of all available valid values after randomization.
Time Frame: 60 minutes post-dose in clinic visits at baseline, and week 0, 3, 7, 12 and Trt Avg
Population: Full analysis set: It consist of all randomized patients who received at least one dose of study medication and contributed sufficient data for at least one efficacy endpoint (Primary variable).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Symbicort BA MDI | Symbicort pMDI | Budesonide
Number analyzed (Participants) | 71 | 71 | 71
Liter
  Baseline | 2.09 (31.46) | 1.97 (27.16) | 2.12 (26.34)
  Week 0 | 2.49 (32.14) | 2.35 (25.97) | 2.28 (27.18)
  Week 3 | 2.52 (31.98) | 2.34 (26.31) | 2.30 (30.22)
  Week 7 | 2.59 (32.17) | 2.35 (27.22) | 2.33 (29.29)
  Week 12 | 2.52 (30.71) | 2.39 (27.31) | 2.30 (28.27)
  Treatment Average | 2.53 (30.57) | 2.37 (26.33) | 2.30 (28.36)
Statistical Analysis 1: Comparison: Symbicort pMDI vs Budesonide; The comparison of Symbicort AC pMDI 2x160/4.5 µg bid with budesonide AC pMDI 2x160 µg bid for post dose FEV1; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA model on the log transformed outcome variable with treatment and country as factor, and log transformed baseline FEV1 (pre-dose) as covariate; Estimated Geometic Mean Ratio = 1.10, 95% CI 2-sided [1.06 to 1.14] — Symbicort AC pMDI 2x160/4.5 µg bid vs Budesonide AC pMDI 2x160 µg bid
Statistical Analysis 2: Comparison: Symbicort BA MDI vs Symbicort pMDI; The comparisons of Symbicort BA MDI 2x160/4.5 µg bid with Symbicort AC pMDI 2x160/4.5 µg bid for post dose FEV1; Test type: Non-Inferiority or Equivalence — Assuming a standard deviation of 0.2 (for pre dose FEV1) on the log-scale and 60 patients/arm, the width of the confidence interval will extend 0.072 from the point estimate on the log-scale. The lower and upper limits of the CI for the ratio of effects will thus be obtained by multiplying the estimated ratio by 0.931 and 1.075, respectively; ANCOVA; [statistical method as in outcome 1, analysis 1]; Estimated Geometric Mean Ratio = 1.01, 95% CI 2-sided [0.97 to 1.05] — The comparisons was used to assess therapeutic equivalence of Symbicort AC pMDI and Symbicort BA MDI. Assay sensitivity was demonstrated before proceeding to assess therapeutic equivalence of the 2 Symbicort products

2. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) - Pre Dose
Description: Descriptive statistics for predose FEV1(L) by visit; Baseline defined as the last pre-dose value prior to 1st dose of randomized therapy. Trt Avg = Mean of all available valid values after randomization.
Time Frame: Pre AM dose in clinic visits at baseline, and week 3, 7, 12 and Trt Avg
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Symbicort BA MDI | Symbicort pMDI | Budesonide
Number analyzed (Participants) | 71 | 71 | 71
Liters
  Baseline | 2.09 (31.46) | 1.97 (27.16) | 2.12 (26.34)
  Week 3 | 2.32 (32.79) | 2.12 (28.29) | 2.22 (31.21)
  Week 7 | 2.40 (32.86) | 2.11 (29.96) | 2.25 (29.01)
  Week 12 | 2.34 (30.84) | 2.17 (31.29) | 2.23 (30.15)
  Average of treatment period | 2.34 (30.15) | 2.15 (29.15) | 2.23 (29.36)
Statistical Analysis 1: Comparison: Symbicort BA MDI vs Symbicort pMDI; The comparisons of Symbicort BA MDI 2x160/4.5 µg bid with Symbicort AC pMDI 2x160/4.5 µg bid, for pre-dose FEV1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; [statistical method as in outcome 1, analysis 1]; Estimated Geometric Mean Ratio = 1.03, 95% CI 2-sided [0.99 to 1.08] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Peak Expiratory Flow
Time Frame: Recorded morning upon rising and evening before sleep for 14 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/Min
Arm/Group | Symbicort BA MDI | Symbicort pMDI | Budesonide
Number analyzed (Participants) | 71 | 71 | 71
L/Min
  Morning Peak expiratory flow (Baseline) | 357.95 (100.59) | 335.70 (102.99) | 360.46 (103.09)
  Evening Peak expiratory flow (Baseline) | 364.61 (103.62) | 347.86 (110.80) | 367.64 (102.73)
  Evening Peak expiratory flow (Treatment Average) | 379.96 (104.72) | 362.99 (112.63) | 348.94 (97.94)
  Morning Peak expiratory flow (Treatment Average) | 376.28 (106.76) | 353.69 (108.72) | 343.59 (98.12)
Statistical Analysis 1: Comparison: Symbicort BA MDI vs Symbicort pMDI; Morning peak expiratory flow (mPEF): Comparing mean changes from baseline to the average of the double-blind treatment period between Symbicort BA MDI 2x160/4.5 μg bid and Symbicort AC pMDI 2x160/4.5 µg bid; Test type: Non-Inferiority or Equivalence — No adjustment were be made for multiplicity for these supportive variables and nominal p-values were reported; p = 0.825, ANCOVA; ANCOVA model includes treatment and country as a factor and baseline value as covariate; Mean Difference (Net) = 1.49, 95% CI 2-sided [-11.81 to 14.80], Standard Error of Mean 6.75 — Secondary efficacy variables were analyzed as continuous data, comparing mean changes from baseline to the average of the double-blind treatment period between treatments. No adjustment were made for multiplicity and nominal p-values were reported
Statistical Analysis 2: Comparison: Symbicort pMDI vs Budesonide; Morning peak expiratory flow (mPEF): Comparing mean changes from baseline to the average of the double-blind treatment period between Symbicort AC pMDI 2x160/4.5 µg bid minus Budesonide AC pMDI 2x160 µg bid; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA model includes treatment and country as a factor and baseline value as covariate; Mean Difference (Net) = 33.52, 95% CI 2-sided [20.11 to 46.93], Standard Error of Mean 6.80 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Symbicort BA MDI vs Symbicort pMDI; Evening peak expiratory flow (ePEF): Comparing mean changes from baseline to the average of the double-blind treatment period between Symbicort BA MDI 2x160/4.5 μg bid and Symbicort AC pMDI 2x160/4.5 µg bid; Test type: Non-Inferiority or Equivalence — No adjustment were made for multiplicity for these supportive variables and nominal p-values were reported; p = 0.810, ANCOVA; ANCOVA model includes treatment and country as a factor and baseline value as covariate; Mean Difference (Net) = 1.48, 95% CI 2-sided [-10.66 to 13.61], Standard Error of Mean 6.15 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Symbicort pMDI vs Budesonide; Evening peak expiratory flow (ePEF): Comparing mean changes from baseline to the average of the double-blind treatment period between Symbicort AC pMDI 2x160/4.5 µg bid and Budesonide AC pMDI 2x160 µg bid; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA model includes treatment and country as a factor and baseline value as covariate; Mean Difference (Net) = 32.25, 95% CI 2-sided [20.01 to 44.49], Standard Error of Mean 6.21 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Asthma Symptoms Score (Total)
Description: The total score is calculated as sum of the morning and evening scores of each day and the treatment period mean score is defined as the mean of all total score recorded during the 12-week treatment period. Trt Avg=Mean total score of double-blind period values.(day/night score ranges from 0 to 3; 0=no asthma symptoms; 3= unable to do normal activities (or to sleep) due to asthma). Higher score represents worse outcome.
Time Frame: Recorded between 6:00 - 11:00 AM from previous 12 hours and 6:00 -11:00 PM from previous 12 hours for 14 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Asthma score on a scale of 0 to 3
Arm/Group | Symbicort BA MDI | Symbicort pMDI | Budesonide
Number analyzed (Participants) | 71 | 71 | 71
Asthma score on a scale of 0 to 3
  Baseline | 2.04 (0.98) | 1.92 (0.72) | 2.12 (0.88)
  Treatment Average (Trt Avg) | 1.68 (1.10) | 1.45 (0.91) | 2.02 (0.96)
Statistical Analysis 1: Comparison: Symbicort BA MDI vs Symbicort pMDI; Comparing mean changes from baseline to the average of the double-blind treatment period between Symbicort BA MDI 2x160/4.5 μg bid and Symbicort AC pMDI 2x160/4.5 µg bid; Test type: Non-Inferiority or Equivalence — No adjustment were made for multiplicity for these supportive variables and nominal p-values were reported; p = 0.272, ANCOVA; ANCOVA model includes treatment and country as a factor and baseline value as covariate; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.10 to 0.35], Standard Error of Mean 0.11

5. Secondary Outcome: Night-time Awakenings Due to Asthma Symptoms(% Awakening-free Nights)
Description: The percentage of days with no awakenings due to asthma. Baseline= Mean % awakening-free nights during run-in period ; Trt Avg=Mean % awakening-free nights during double-blind period.
Time Frame: Recorded 6:00 - 11:00 AM for 14 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days with no awakenings
Arm/Group | Symbicort BA MDI | Symbicort pMDI | Budesonide
Number analyzed (Participants) | 71 | 71 | 71
Percentage of days with no awakenings
  Baseline | 78.54 (28.97) | 78.76 (29.76) | 81.59 (25.32)
  Treatment Average (Trt Avg) | 83.73 (30.90) | 89.93 (21.40) | 84.62 (26.31)
Statistical Analysis 1: Comparison: Symbicort BA MDI vs Symbicort pMDI; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — No adjustment were made for multiplicity for these supportive variables and nominal p-values were reported; p = 0.025, ANCOVA; ANCOVA model includes treatment and country as a factor and baseline value as covariate; Mean Difference (Net) = -6.10, 95% CI 2-sided [-11.41 to -0.79], Standard Error of Mean 2.69

6. Secondary Outcome: Use of Rescue Medication Day and Night (Total Daily Rescue Medication Use)
Description: Total daily rescue medication use is calculated as the sum of morning and evening use each day and averaged over the 12 weeks treatment periods to calculate the treatment period mean. Baseline= Mean rescue medication used during run-in period ; Trt Avg=Mean rescue medication used during double-blind period.
Time Frame: Recorded between 6:00 - 11:00 AM from previous 12 hours and 6:00 -11:00 PM from previous 12 hours for 14 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Inhalations/24 hrs
Arm/Group | Symbicort BA MDI | Symbicort pMDI | Budesonide
Number analyzed (Participants) | 71 | 71 | 71
Inhalations/24 hrs
  Baseline | 2.55 (2.48) | 2.19 (1.75) | 2.65 (2.36)
  Treatment Average (Trt Avg) | 1.81 (2.67) | 1.26 (1.60) | 2.34 (2.38)
Statistical Analysis 1: Comparison: Symbicort BA MDI vs Symbicort pMDI; Comparing mean changes from baseline to the average of the double-blind treatment period between BAI Symbicort BA MDI 2x160/4.5 μg bid and pMDI Symbicort AC pMDI 2x160/4.5 µg bid; Test type: Non-Inferiority or Equivalence — No adjustment were made for multiplicity for these supportive variables and nominal p-values were reported; p = 0.258, ANCOVA; ANCOVA model includes treatment and country as a factor and baseline value as covariate; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.19 to 0.71], Standard Error of Mean 0.23

ADVERSE EVENTS:
Description: 'Number of participants in the safety analysis set is (71 for all the group)as 1 patients from the Budesonide group has not taken any dose of the IP, so not included in the Safety population'
Arm/Group | Budesonide | Symbicort BA MDI | Symbicort pMDI
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71 | 1/71
Other Adverse Events (participants affected / at risk) | 3/71 | 2/71 | 7/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide (N=71) | Symbicort BA MDI (N=71) | Symbicort pMDI (N=71)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide (N=71) | Symbicort BA MDI (N=71) | Symbicort pMDI (N=71)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2) | 7 (7)

LIMITATIONS AND CAVEATS:
No. of participants in the safety analysis set is (71 for all the group) as 1 patients from the Budesonide group has not taken any dose of the IP, so not included in the Safety population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than less than or equal to 180 days from the date of AZ's request to allow for the filing of a patent app or the taking of such measures as AZ deems appropriate to establish and preserve its proprietary rights in teh material being submitted.